CLINICAL TRIAL: NCT00632788
Title: The Influence of Acute Myocardial Infarction Checklist on the Door-to-Balloon Time in Patients Suffering From Acute ST-Elevation Myocardial Infarction
Brief Title: The Influence of Acute Myocardial Infarction Checklist on the Door-to-Balloon Time
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Lai, Chao-Lun, Far Eastern Memorial Hospital
Other Study IDs: 97005
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-01

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; catheterization; angioplasty; door-to-balloon time
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intervention group: patients presented with acute ST-elevation myocardial infarction and received emergency cardiac catheterization between March 1, 2007 and Oct. 31, 2007
  Interventions: Other: acute myocardial infarction checklist
- control group: patients presented with acute ST-elevation myocardial infarction and received emergency cardiac catheterization between April 1, 2006 and Feb. 28, 2007

INTERVENTIONS:
Other: acute myocardial infarction checklist — For every patient fulfilling the criteria of enrollment, an acute myocardial infarction checklist was incorporated into the patient's medical records at emergency department immediately after a diagnosis of acute ST-elevation myocardial infarction was made. All the time sequences concerning different managements at different locations were recorded by nurses and/or physicians as instructions on the checklist.
  Groups: intervention group

SUMMARY:
This study was designed to investigate the influence of the acute myocardial infarction checklist on the door-to-balloon time in patients suffering from acute STEMI at Far Eastern Memorial Hospital

ELIGIBILITY:
Inclusion Criteria:

* all patients who presented to the emergency department of Far Eastern Memorial Hospital within 12 hours of the onset of ischemic chest pain
* patients with diagnostic criteria of acute ST-elevation myocardial infarction on electrocardiogram, e.g. at least 0.1 mV in two or more contiguous electrocardiographic leads or a new onset of bundle branch block
* patients were preparing for emergency cardiac catheterization

Exclusion Criteria:

* patients who did not fulfill the diagnostic criteria of acute myocardial infarction on electrocardiogram
* patients who were not eligible for cardiac catheterization
* patients who refused cardiac catheterization
* patients who suffered from acute myocardial infarction after admission to ward or intensive care unit for any reason
* patients who had an ambiguous diagnosis that the decision of emergency cardiac catheterization was made after admission to ward or intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diagnostic criteria of acute ST-elevation myocardial infarction who were preparing for emergency cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
median door-to-balloon time | at cath. lab

SECONDARY OUTCOMES:
in-hospital mortality | at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Lun Lai, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lai CL, Fan CM, Liao PC, Tsai KC, Yang CY, Chu SH, Chien KL. Impact of an audit program and other factors on door-to-balloon times in acute ST-elevation myocardial infarction patients destined for primary coronary intervention. Acad Emerg Med. 2009 Apr;16(4):333-42. doi: 10.1111/j.1553-2712.2009.00372.x. PMID 19456296